CLINICAL TRIAL: NCT06417112
Title: Can Left Atrial Strain Measurements, and Correlating Changes in Left Atrium Area and Volume Size, be Used as an Early Predictor of Atrial Fibrillation?
Brief Title: Left Atrial Strain Values as an Early Predictor of Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Hywel Dda Health Board (Other)
Responsible Party: Principal Investigator, Lucy Hwozdyk, Trainee Clinical Cardiac Scientist, Hywel Dda Health Board
Other Study IDs: 324893
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Hypertension
Keywords: atrial fibrillation; hypertension; LA size; LA strain; LA reservoir strain; LA conduit strain; LA contractile strain
MeSH Terms: conditions — Atrial Fibrillation; Hypertension | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal sinus rhythm and normotensive: All participants are in normal sinus rhythm at the time of the transthoracic echocardiogram and no previous history of atrial fibrillation.
  All participants have blood pressure measurements within normal limits and are not prescribed anti-hypertensive medication.
  Interventions: Diagnostic Test: Transthoracic Echocardiogram
- Normal sinus rhythm and hypertensive: All participants are in normal sinus rhythm at the time of the transthoracic echocardiogram and no previous history of atrial fibrillation.
  All participants are known to have raised blood pressure measurements previously and are receiving anti-hypertensive medication.
  Interventions: Diagnostic Test: Transthoracic Echocardiogram
- Known atrial fibrillation: All participants are known to have a history of atrial fibrillation (paroxysmal, persistent or permanent).
  Interventions: Diagnostic Test: Transthoracic Echocardiogram

INTERVENTIONS:
Diagnostic Test: Transthoracic Echocardiogram — All participants have been referred for a transthoracic echocardiogram by a clinician.

SUMMARY:
Atrial fibrillation (AF) is the most common type of abnormal heart rhythm. This occurs as the chambers of the heart pump irregularly, often resulting in a fast heart rate and symptoms of irregular pounding and fluttering. There are many risk factors predisposing to AF, however, the cause cannot always be easily determined. Additionally, not all AF patients experience symptoms and consequently, this abnormal rhythm may go undetected and may be discovered accidentally. This is detrimental to patients, as untreated AF patients are at an increased risk of stroke.

Patients that are suspected of having AF are referred for an ultrasound scan of the heart (echocardiogram). It is expected to see structural changes to the heart's chambers. However, structural and electrical changes of the heart may be the cause of AF but may also be a result of AF, resulting in a chicken and egg situation. It may be possible that a different type of measurement can be used during an echocardiogram to detect subtle changes in heart muscle patterns. This measurement may then serve to be an early predictor of AF. This would be determined by comparing the patterns in patients with a normal, regular rhythm to those with AF.

Potential candidates are initially screened based on their echocardiogram referral. If deemed suitable for this study, the study process is explained to the patient and written informed consent is invited and received. The echocardiogram will be performed as normal with a focus on the area and volume measurements taken of one of the top chambers of the heart. An additional measurement will be taken to observe any subtle changes in the arrangement of heart cells within this same heart chamber. These measurements can be compared to each other to establish any relationship as well as compared to patients with and without AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most prevalent type of arrhythmia within an adult population and is characterised by disorganised, chaotic, electrical activity and thus, ineffective atrial contraction causing irregular ventricular contraction. AF can be categorised into three different groups: paroxysmal, persistent and permanent. The prevalence of AF increases with age and is associated with a range of risk factors including: hypertension, obesity and alcohol consumption. There is a plethora of both cardiac and non-cardiac causes of AF and the cause is not always clear for each patient. Furthermore, causes of AF can also present as the by-product of AF, this increases the difficulty in determining the individual patient's cause of onset. A diagnosis of AF can be incidental as not all patients are symptomatic. If AF goes undetected, this puts the patient at an increased risk of blood clot formation and stroke.

Patients suspected of having AF are routinely referred for a transthoracic echocardiogram (TTE). It is common for AF patients to have a dilated left atrium (LA). This can be visually confirmed, and the LA area and volume can be measured during a TTE. LA strain measurements are not routinely measured during TTEs but may be able to detect subtle changes in longitudinal strain patterns of the myocardium. By comparing the strain patterns in patients with normal sinus rhythm (control) to those with AF, a scale can be created to suggest and predict whether a patient is likely to develop AF in the future based on these subtle changes before any changes in LA size occur. Furthermore, this can then be further developed to determine whether there are any significant differences in strain patterns between the three AF groups.

Objectives:

To determine whether there is a significant difference in atrial strain values between patients that are in normal sinus rhythm (NSR, control group) to patients that are known to have atrial fibrillation (disease group). A disease-control group of controlled hypertensive patients in NSR will also be utilised as hypertension is a known risk factor for atrial fibrillation.

Providing that there is a significant difference in the values between NSR and AF patients, a further comparison will be conducted on patients in different type of AF: paroxysmal AF, persistent AF and permanent AF to determine if there is a deterioration in atrial strain values within AF patients.

Left atrial area and volume size will also be measured in all patients and this can then be compared to atrial strain values.

ELIGIBILITY:
Inclusion Criteria:

* Criterion 1: subjects will be included in the study if they are within one of the following groups:

  * Known to be in normal sinus rhythm, are normotensive and have no underlying health problems.
  * Known to be in normal sinus rhythm and have controlled hypertension. This must have been diagnosed by a healthcare professional and the patient should be taking appropriate antihypertensive medication.
  * Known to have chronic atrial fibrillation (persistent or permanent AF). This must have been diagnosed by a healthcare professional and the patient should be appropriately anticoagulated.
* Criterion 2: subjects should ideally be ≥ 50 years, but subjects will be age matched across all three groups.
* Criterion 3: patients should have an EF ≥ 50%.
* Criterion 4: good quality TTE images.
* Criterion 5: No valvular pathologies. o Patients with AF that have < moderate valvular pathologies may be considered (as per the British Society of Echocardiography Guidelines).

Exclusion Criteria:

* Criterion 1: subjects with any valvular pathologies in the control and disease- control groups.
* Criterion 2: subjects with AF that have ≥ moderate valvular pathologies (as per the British Society of Echocardiography Guidelines).
* Criterion 3: subjects with an EF < 50%.
* Criterion 4: subjects < 50 years old.
* Criterion 5: poor quality TTE images.
* Criterion 6: inability to provide informed consent.
* Criterion 7: permanent atrial / ventricular pacing.
* Criterion 8: previous cardiac surgery.
* Criterion 9: unsatisfactory tracking of the LA endocardial border.
* Criterion 10: patients unwilling to have their results potentially published.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To be included, patients had to be categorised into one of the following categories: normal sinus rhythm and normotensive, normal sinus rhythm and hypertensive, or known chronic atrial fibrillation. Additionally, all eligible patients had to conform to the aforementioned inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Left atrial strain values | Baseline
  Taking measurements to assess left atrial strain from two different views (A4C & A2C) as well as biplane measurements for reservoir, contractile and conduit LA strain.
LA volume size | Baseline
  Taking measurements to assess left atrial volume from two different views (A4C & A2C) as well as biplane measurements.
LA area size | Baseline
  Taking measurements to assess left atrial area from A4C view.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Hwozdyk, Principal Investigator — Hywel Dda University Health Board
Locations (1):
- Lucy Hwozdyk, Haverfordwest, Pembrokeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
All participant data has been pseudo-anonymised, this prevents any information from being able to be used to trace back to individual participants. Anonymised data may be able to be shared with other researchers rather than the mean data used in the data analyses.

REFERENCES:
- [Result] Alhakak AS, Biering-Sorensen SR, Mogelvang R, Modin D, Jensen GB, Schnohr P, Iversen AZ, Svendsen JH, Jespersen T, Gislason G, Biering-Sorensen T. Usefulness of left atrial strain for predicting incident atrial fibrillation and ischaemic stroke in the general population. Eur Heart J Cardiovasc Imaging. 2022 Feb 22;23(3):363-371. doi: 10.1093/ehjci/jeaa287. PMID 33175146
- [Result] Beyls C, Hermida A, Bohbot Y, Martin N, Viart C, Boisgard S, Daumin C, Huette P, Dupont H, Abou-Arab O, Mahjoub Y. Automated left atrial strain analysis for predicting atrial fibrillation in severe COVID-19 pneumonia: a prospective study. Ann Intensive Care. 2021 Dec 7;11(1):168. doi: 10.1186/s13613-021-00955-w. PMID 34874509
- [Result] Choi HM, Yoon YE, Oh IY, Cho Y, Cho GY. Global Left Atrial Strain as a Predictor of Silent Atrial Fibrillation Following Dual Chamber Cardiac Implantable Electronic Device Implantation. JACC Cardiovasc Imaging. 2018 Oct;11(10):1537-1539. doi: 10.1016/j.jcmg.2017.12.013. Epub 2018 Feb 14. No abstract available. PMID 29454782
- [Result] Gan GCH, Ferkh A, Boyd A, Thomas L. Left atrial function: evaluation by strain analysis. Cardiovasc Diagn Ther. 2018 Feb;8(1):29-46. doi: 10.21037/cdt.2017.06.08. PMID 29541609
- [Result] Guo C, Liu J, Zhao S, Teng Y, Shen L. Decreased left atrial strain parameters are correlated with prolonged total atrial conduction time in lone atrial fibrillation. Int J Cardiovasc Imaging. 2016 Jul;32(7):1053-61. doi: 10.1007/s10554-016-0875-3. Epub 2016 Apr 13. PMID 27076225
- [Result] Hauser R, Nielsen AB, Skaarup KG, Lassen MCH, Duus LS, Johansen ND, Sengelov M, Marott JL, Jensen G, Schnohr P, Sogaard P, Mogelvang R, Biering-Sorensen T. Left atrial strain predicts incident atrial fibrillation in the general population: the Copenhagen City Heart Study. Eur Heart J Cardiovasc Imaging. 2021 Dec 18;23(1):52-60. doi: 10.1093/ehjci/jeab202. PMID 34632488
- [Result] Her AY, Kim JY, Kim YH, Choi EY, Min PK, Yoon YW, Lee BK, Hong BK, Rim SJ, Kwon HM. Left atrial strain assessed by speckle tracking imaging is related to new-onset atrial fibrillation after coronary artery bypass grafting. Can J Cardiol. 2013 Mar;29(3):377-83. doi: 10.1016/j.cjca.2012.06.006. Epub 2012 Aug 15. PMID 22902158
- [Result] Hsu PC, Lee WH, Chu CY, Lee HH, Lee CS, Yen HW, Lin TH, Voon WC, Lai WT, Sheu SH, Su HM. Prognostic role of left atrial strain and its combination index with transmitral E-wave velocity in patients with atrial fibrillation. Sci Rep. 2016 Feb 1;6:17318. doi: 10.1038/srep17318. PMID 26833057
- [Result] Jarasunas J, Aidietis A, Aidietiene S. Left atrial strain - an early marker of left ventricular diastolic dysfunction in patients with hypertension and paroxysmal atrial fibrillation. Cardiovasc Ultrasound. 2018 Oct 31;16(1):29. doi: 10.1186/s12947-018-0147-6. PMID 30382851
- [Result] Ma XX, Zhang YL, Hu B, Zhu MR, Jiang WJ, Wang M, Zheng DY, Xue XP. The usefulness of global left atrial strain for predicting atrial fibrillation recurrence after catheter ablation in patients with persistent and paroxysmal atrial fibrillation. Arch Cardiovasc Dis. 2017 Aug-Sep;110(8-9):447-455. doi: 10.1016/j.acvd.2016.11.005. Epub 2017 May 18. PMID 28528995
- [Result] Markides V, Schilling RJ. Atrial fibrillation: classification, pathophysiology, mechanisms and drug treatment. Heart. 2003 Aug;89(8):939-43. doi: 10.1136/heart.89.8.939. No abstract available. PMID 12860883
- [Result] Mochizuki A, Yuda S, Fujito T, Kawamukai M, Muranaka A, Nagahara D, Shimoshige S, Hashimoto A, Miura T. Left atrial strain assessed by three-dimensional speckle tracking echocardiography predicts atrial fibrillation recurrence after catheter ablation in patients with paroxysmal atrial fibrillation. J Echocardiogr. 2017 Jun;15(2):79-87. doi: 10.1007/s12574-017-0329-5. Epub 2017 Feb 2. PMID 28155065
- [Result] Motoki H, Negishi K, Kusunose K, Popovic ZB, Bhargava M, Wazni OM, Saliba WI, Chung MK, Marwick TH, Klein AL. Global left atrial strain in the prediction of sinus rhythm maintenance after catheter ablation for atrial fibrillation. J Am Soc Echocardiogr. 2014 Nov;27(11):1184-92. doi: 10.1016/j.echo.2014.08.017. Epub 2014 Sep 23. PMID 25260436
- [Result] Olsen FJ, Christensen LM, Krieger DW, Hojberg S, Host N, Karlsen FM, Svendsen JH, Christensen H, Biering-Sorensen T. Relationship between left atrial strain, diastolic dysfunction and subclinical atrial fibrillation in patients with cryptogenic stroke: the SURPRISE echo substudy. Int J Cardiovasc Imaging. 2020 Jan;36(1):79-89. doi: 10.1007/s10554-019-01700-y. Epub 2019 Oct 8. PMID 31595399
- [Result] Pagola J, Juega J, Francisco-Pascual J, Bustamante A, Penalba A, Pala E, Rodriguez M, De Lera-Alfonso M, Arenillas JF, Cabezas JA, Moniche F, de Torres R, Montaner J, Gonzalez-Alujas T, Alvarez-Sabin J, Molina CA; Crypto-AF study group. Predicting Atrial Fibrillation with High Risk of Embolization with Atrial Strain and NT-proBNP. Transl Stroke Res. 2021 Oct;12(5):735-741. doi: 10.1007/s12975-020-00873-2. Epub 2020 Nov 13. PMID 33184686
- [Result] Park JJ, Park JH, Hwang IC, Park JB, Cho GY, Marwick TH. Left Atrial Strain as a Predictor of New-Onset Atrial Fibrillation in Patients With Heart Failure. JACC Cardiovasc Imaging. 2020 Oct;13(10):2071-2081. doi: 10.1016/j.jcmg.2020.04.031. Epub 2020 Jul 15. PMID 32682715
- [Result] Parwani AS, Morris DA, Blaschke F, Huemer M, Pieske B, Haverkamp W, Boldt LH. Left atrial strain predicts recurrence of atrial arrhythmias after catheter ablation of persistent atrial fibrillation. Open Heart. 2017 Apr 28;4(1):e000572. doi: 10.1136/openhrt-2016-000572. eCollection 2017. PMID 28674624
- [Result] Pathan F, Sivaraj E, Negishi K, Rafiudeen R, Pathan S, D'Elia N, Galligan J, Neilson S, Fonseca R, Marwick TH. Use of Atrial Strain to Predict Atrial Fibrillation After Cerebral Ischemia. JACC Cardiovasc Imaging. 2018 Nov;11(11):1557-1565. doi: 10.1016/j.jcmg.2017.07.027. Epub 2017 Nov 15. PMID 29153561
- [Result] Pessoa-Amorim G, Mancio J, Vouga L, Ribeiro J, Gama V, Bettencourt N, Fontes-Carvalho R. Impaired Left Atrial Strain as a Predictor of New-onset Atrial Fibrillation After Aortic Valve Replacement Independently of Left Atrial Size. Rev Esp Cardiol (Engl Ed). 2018 Jun;71(6):466-476. doi: 10.1016/j.rec.2017.10.005. Epub 2017 Nov 14. English, Spanish. PMID 29146482
- [Result] Petre I, Onciul S, Iancovici S, Zamfir D, Stoian M, Scarlatescu A, Diaconeasa A, Acatrinei C, Dorobantu M. Left Atrial Strain for Predicting Atrial Fibrillation Onset in Hypertensive Patients. High Blood Press Cardiovasc Prev. 2019 Aug;26(4):331-337. doi: 10.1007/s40292-019-00326-4. Epub 2019 Jul 15. PMID 31309456
- [Result] Rasmussen SMA, Olsen FJ, Jorgensen PG, Fritz-Hansen T, Jespersen T, Gislason G, Biering-Sorensen T. Utility of left atrial strain for predicting atrial fibrillation following ischemic stroke. Int J Cardiovasc Imaging. 2019 Sep;35(9):1605-1613. doi: 10.1007/s10554-019-01601-0. Epub 2019 Apr 26. PMID 31028567
- [Result] Shaikh AY, Maan A, Khan UA, Aurigemma GP, Hill JC, Kane JL, Tighe DA, Mick E, McManus DD. Speckle echocardiographic left atrial strain and stiffness index as predictors of maintenance of sinus rhythm after cardioversion for atrial fibrillation: a prospective study. Cardiovasc Ultrasound. 2012 Dec 3;10:48. doi: 10.1186/1476-7120-10-48. PMID 23199055
- [Result] Shin DG, Kang MK, Han D, Choi S, Cho JR, Lee N. Enlarged left atrium and decreased left atrial strain are associated with atrial fibrillation in patients with hyperthyroidism irrespective of conventional risk factors. Int J Cardiovasc Imaging. 2022 Mar;38(3):613-620. doi: 10.1007/s10554-021-02450-6. Epub 2021 Oct 27. PMID 34705162
- [Result] Singh A, El Hangouche N, McGee K, Gong FF, Lentz R, Feinglass J, Akhter N. Utilizing left atrial strain to identify patients at risk for atrial fibrillation on ibrutinib. Echocardiography. 2021 Jan;38(1):81-88. doi: 10.1111/echo.14946. Epub 2020 Dec 7. PMID 33594858
- [Result] Staerk L, Sherer JA, Ko D, Benjamin EJ, Helm RH. Atrial Fibrillation: Epidemiology, Pathophysiology, and Clinical Outcomes. Circ Res. 2017 Apr 28;120(9):1501-1517. doi: 10.1161/CIRCRESAHA.117.309732. PMID 28450367
- [Result] Svartstein AW, Lassen MH, Skaarup KG, Grove GL, Vyff F, Ravnkilde K, Pedersen S, Galatius S, Modin D, Biering-Sorensen T. Predictive value of left atrial strain in relation to atrial fibrillation following acute myocardial infarction. Int J Cardiol. 2022 Oct 1;364:52-59. doi: 10.1016/j.ijcard.2022.05.026. Epub 2022 May 14. PMID 35577164
- [Result] Uzieblo-Zyczkowska B, Krzesinski P, Jurek A, Krzyzanowski K, Kiliszek M. Correlations between left atrial strain and left atrial pressures values in patients undergoing atrial fibrillation ablation. Kardiol Pol. 2021;79(11):1223-1230. doi: 10.33963/KP.a2021.0113. Epub 2021 Oct 2. PMID 34599496
- [Result] van de Vegte YJ, Siland JE, Rienstra M, van der Harst P. Atrial fibrillation and left atrial size and function: a Mendelian randomization study. Sci Rep. 2021 Apr 19;11(1):8431. doi: 10.1038/s41598-021-87859-8. PMID 33875748
- [Result] von Roeder M, Rommel KP, Kowallick JT, Blazek S, Besler C, Fengler K, Lotz J, Hasenfuss G, Lucke C, Gutberlet M, Schuler G, Schuster A, Lurz P. Influence of Left Atrial Function on Exercise Capacity and Left Ventricular Function in Patients With Heart Failure and Preserved Ejection Fraction. Circ Cardiovasc Imaging. 2017 Apr;10(4):e005467. doi: 10.1161/CIRCIMAGING.116.005467. PMID 28360259
- [Result] Wyndham CR. Atrial fibrillation: the most common arrhythmia. Tex Heart Inst J. 2000;27(3):257-67. PMID 11093410
- [Result] Yasuda R, Murata M, Roberts R, Tokuda H, Minakata Y, Suzuki K, Tsuruta H, Kimura T, Nishiyama N, Fukumoto K, Aizawa Y, Tanimoto K, Takatsuki S, Abe T, Fukuda K. Left atrial strain is a powerful predictor of atrial fibrillation recurrence after catheter ablation: study of a heterogeneous population with sinus rhythm or atrial fibrillation. Eur Heart J Cardiovasc Imaging. 2015 Sep;16(9):1008-14. doi: 10.1093/ehjci/jev028. Epub 2015 Mar 6. PMID 25750193
- See also: Incremental value of left atrial strain to predict atrial fibrillation recurrence after cryoballoon ablation — https://researchportal.vub.be/en/publications/incremental-value-of-left-atrial-strain-to-predict-atrial-fibrill

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT06417112/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT06417112/ICF_001.pdf